CLINICAL TRIAL: NCT01631630
Title: Role of Proinflammatory Signaling in Alcohol Craving
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was closed to recruitment due to feasibility problems.
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 120143; 12-AA-0143 (Other: NIH)
Record Dates: First submitted 2012-06-27; First posted 2012-06-29 (Estimated); Results first posted 2016-12-15 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-01

CONDITIONS: Alcohol Dependence; Alcohol Drinking; Stress; Alcohol-Related Disorders
Keywords: Alcohol; Alcohol Dependence; Alcohol Use; Nicotine Dependence; Nicotine
MeSH Terms: conditions — Alcoholism; Alcohol Drinking; Alcohol-Related Disorders; Tobacco Use Disorder | interventions — Pioglitazone; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pioglitazone (Experimental): Subjects received pioglitazone, 15mg/day for 3 days; 30mg day for 3 days; 45mg/day thereafter, for a minimum total of 13 days
  Interventions: Drug: Pioglitazone
- Placebo (Placebo Comparator): Subjects received placebo on a similar dosing schedule, for a minimum total of 13 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pioglitazone — Pioglitazone is a thiazolidinedione antidiabetic. It works by lowering blood sugar by making the cells of the body more sensitive to the action of insulin.
  Other Names: Actos
  Arms: Pioglitazone
Drug: Placebo — Placebo is an inactive tablet design to look exactly like pioglitazone
  Other Names: Sugar Pill
  Arms: Placebo

SUMMARY:
Background:

- Drinking too much alcohol can injure cells in the body. Inflammation is the body s reaction to injured cells. Studies show that inflammation can cause cravings for alcohol. Researchers want to see if pioglitazone, a drug that decreases inflammation, can reduce alcohol craving. If so, it might help develop new ways to help alcoholics with craving.

Objectives:

- To see if pioglitazone can reduce alcohol craving.

Eligibility:

- Adults between 21 and 65 years of age who are alcoholic and have been drinking within the past month.

Design:

* Participants will be screened with a physical exam and medical history. Blood samples will also be collected.
* All participants will have inpatient treatment at the National Institutes of Health Clinical Center for the 5 weeks of the study. They will have standard treatment for alcoholism during their inpatient stay.
* Half of the people in this study will have pioglitazone. The other half will have a placebo.
* Participants will have different studies during their stay. These studies will include the following:
* Personalized audio recordings of stressful, alcohol-related, and neutral events to monitor mood
* Imaging studies to test alcohol cravings
* Questionnaires about mood and alcohol cravings
* Lumbar puncture to collect spinal fluid
* Inflammation test to see if the study drug can block alcohol cravings
* After the end of the 5-week study, all participants will be offered follow-up outpatient care through the Clinical Center, or referral to outside treatment.

DETAILED DESCRIPTION:
Objective: The objective of the present study is to evaluate the role of proinflammatory signaling in alcohol craving. The peroxisome proliferator-activated receptor y (PPARy) agonist pioglitazone, which modulates glial activity, will be used as an experimental treatment. Guided imagery auditory scripts will be used as an established set of stimuli to induce craving. Low dose lipopolysaccharide (LPS) administration which activates proinflammatory signaling will be used as a novel challenge, and evaluated for its ability to provoke alcohol craving. If LPS in fact induces alcohol craving, the present design will allow evaluation of whether pioglitazone can inhibit this response.

Study population: Up to 60 subjects will be recruited for a target accrual of 50 completers. Subjects will be aged 21-65 years, with alcohol dependence as their primary complaint, and without other serious medical or psychiatric conditions. They will be admitted to the NIAAA research inpatient unit at the NIH Clinical Research Center (CRC) through one of the screening protocols (05-AA-0121 Assessment and Treatment of People with Alcohol Drinking Problems ) or 14-AA-0181 "Unit and Clinic Evaluations, Screening, Assessment, and Management") which provides basic assessments and standard withdrawal treatment if needed.

Design: Following inclusion, subjects will undergo interviews for construction of guided imagery scripts, and these scripts will subsequently be used as stress-, alcohol- or neutral condition associated stimuli. Subjects will be randomized to pioglitazone (n=25; final dose: 45mg/daily) or identically looking placebo (n=25). Following at least two weeks of treatment, subjects will undergo three sessions of guided imagery, on separate days and in a counter-balanced order, exposing them to the personalized stress-, alcohol- or neutral condition associated auditory scripts, respectively. During the final week, subjects will undergo two challenge sessions, a minimum of five days apart, with lipopolysaccharide (LPS) or placebo, in counterbalanced order.

Outcome measures: Subjective ratings of mood, anxiety and craving will be obtained twice weekly throughout the study. During the challenge sessions that utilize psychological stimuli or LPS, subjective ratings of craving for alcohol, as well as ratings of negative emotions will be obtained. Lumbar puncture will be performed and cerebrospinal fluid (CSF) obtained to determine the effect of pioglitazone on levels of proinflammatory cytokines. Neuroendocrine, psychological and physiological measures will be collected for exploratory purposes. An fMRI scan will be obtained to evaluate the effect of pioglitazone on BOLD signal in response to emotionally salient visual cues.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Diagnostic and Statistical Manual (DSM)-IV diagnosis of alcohol dependence on Structured Clinical Interview for DSM Diagnosis (SCID) alcohol problems as primary complaint among substance use disorders, and alcohol use within the last month.
  2. Age 21 65
  3. Right handed
  4. For women:

     1. post-menopausal or surgically sterile (tubal ligation or hysterectomy); or
     2. if sexually active with a male partner and able to get pregnant, documented agreement to use an effective form of birth control. Acceptable forms of contraception for this study include: hormonal contraceptives (birth-control pills, injectable hormones, vaginal-ring hormones); intrauterine device (IUD); diaphragm with spermicide; condom with spermicide.

EXCLUSION CRITERIA:

1. Any medical illness that in the view of the investigators would compromise participation in research, as determined by medical history, physical examination, laboratory tests (see details under Screening measures below), including, but not limited to:

   1. Diabetes mellitus Type I or Type II
   2. Past or current diagnosis of congestive heart failure
   3. Signs and symptoms suggestive of congestive heart failure
   4. Cardiovascular disease (e.g., history of congenital heart defect, heart disease, symptomatic coronary-artery disease, heart attack, clinically significant arrhythmia, etc.)
   5. Cerebrovascular disease
   6. Infection, autoimmune disease, or fever of unknown origin
   7. Unexplained history of syncope
   8. History of seizures, except for febrile seizures during childhood
   9. History of head injury with loss of consciousness of more than 30 minutes or with postconcussive sequelae lasting more than two days, regardless of loss of consciousness
   10. Chronic renal failure as estimated by glomerular filtration rate (GFR) <60 milliliters per minute 1.73 per Square
   11. HIV infection
   12. Active bladder cancer, history of bladder cancer, or persistent hematuria
   13. Allergy, hypersensitivity, or intolerance to pioglitazone, other thiazolidinediones, or the metabolites of any of those drugs (determined by medical history)
   14. Pregnancy or breastfeeding (urine pregnancy test; self-report)
   15. Diabetes medications (e.g., sulfonylureas, metformin, insulin, etc.)
   16. Contraindicated or strongly interacting medications: Gemfibrozil (inhibitor of CYP2C8) and rifampin (inducer of CYP2C8), atorvastatin, ketoconazole, nifedipine
   17. Any ongoing, or regular use of central nervous system (CNS) active medications within the last week (fluoxetine: last 4 weeks), with the exception of withdrawal medication, obtained according to the NIAAA clinical guidelines if needed
   18. Use of docosahexaenoic acid (DHA) dietary supplements, or consumption of oily fish >3 times per week (because of effects of DHA on inflammatory parameters)
   19. History of Rhabdomyolysis
2. Psychiatric history:

   1. Cognitive impairment severe enough to preclude informed consent or valid responses on questionnaires, as established by clinical exam, in questionable cases aided by a Mini Mental State Examination (with a score of <21, indicating more than mild cognitive impairment, being exclusionary)
   2. Current diagnosis of schizophrenia or any other DSM-IV psychotic disorder, bipolar disorder, or major depressive disorder, in each case as established by clinical evaluation and SCID.
3. Substance use disorders:

   1. Current alcohol intoxication on breathalyzer test or positive urine drug screen on enrollment
   2. Current dependence on drugs other than alcohol or nicotine, as established by SCID interview
4. Inability or unwillingness to participate in an fMRI scan, including

   1. Presence of ferromagnetic objects in the body that are contraindicated for MRI of the head (pacemakers or other implanted electrical devices, brain stimulators, some types of dental implants, aneurysm clips, metallic prostheses, permanent eyeliner, implanted delivery pump, or shrapnel fragments) or fear of enclosed spaces. Eligibility will be determined by a MRI Safety Screening Questionnaire and verified, if necessary, by a physician.
   2. Subjects that cannot lie comfortably flat on their back for up to 2 hours in the MRI scanner.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-05; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Diazgranados, M.D., Principal Investigator — National Institute on Alcohol Abuse and Alcoholism (NIAAA)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Capuron L, Miller AH. Immune system to brain signaling: neuropsychopharmacological implications. Pharmacol Ther. 2011 May;130(2):226-38. doi: 10.1016/j.pharmthera.2011.01.014. Epub 2011 Feb 17. PMID 21334376
- [Background] Crews FT, Zou J, Qin L. Induction of innate immune genes in brain create the neurobiology of addiction. Brain Behav Immun. 2011 Jun;25 Suppl 1(Suppl 1):S4-S12. doi: 10.1016/j.bbi.2011.03.003. Epub 2011 Mar 21. PMID 21402143
- [Background] Dantzer R, Kelley KW. Twenty years of research on cytokine-induced sickness behavior. Brain Behav Immun. 2007 Feb;21(2):153-60. doi: 10.1016/j.bbi.2006.09.006. Epub 2006 Nov 7. PMID 17088043
- [Derived] Schwandt ML, Diazgranados N, Umhau JC, Kwako LE, George DT, Heilig M. PPARgamma activation by pioglitazone does not suppress cravings for alcohol, and is associated with a risk of myopathy in treatment seeking alcohol dependent patients: a randomized controlled proof of principle study. Psychopharmacology (Berl). 2020 Aug;237(8):2367-2380. doi: 10.1007/s00213-020-05540-w. Epub 2020 May 22. PMID 32445052
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2012-AA-0143.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Subjects received placebo on a similar dosing schedule as pioglitazone, for a minimum total of 13 days
Period: Overall Study
Arm/Group | Pioglitazone | Placebo
Started | 8 | 8
Completed | 5 | 8
Not Completed | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pioglitazone | Placebo | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants]
  LTE18 | 0 | 0 | 0
  BTWN | 8 | 8 | 16
  GTE65 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 8 | 7 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 8 | 16
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Hawaiian | 0 | 0 | 0
  Black | 5 | 4 | 9
  White | 2 | 3 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Alcohol Craving in Response to the Alcohol Cue Script
Description: Alcohol craving was measured using the Alcohol Urges Questionnaire (AUQ). The AUQ is an 8-item self-administered instrument that assesses craving for alcohol among alcohol users in the current context (i.e., right now). The score ranges from 8 (lowest craving value) to 56 (highest craving value).
Time Frame: 15 minutes prior to the beginning of script presentation, which occurred on Day 21, 22, or 23 of the treatment period
Population: The analyses included only those subjects who completed all three script types (neutral, alcohol, stress)
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 6 | 8
Units on a scale | 13.7505 (2.3136) | 8.1871 (1.9853)

2. Primary Outcome: Alcohol Craving in Response to the Alcohol Cue Script
Description: as for outcome 1
Time Frame: 5 minutes after the beginning of script presentation, which occurred on Day 21, 22, or 23 of the treatment period
Population: The analyses included only those subjects who completed all three script types (neutral, alcohol, stress)
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 6 | 8
Units on a scale | 20.5838 (2.3136) | 9.6871 (1.9853)

3. Primary Outcome: Alcohol Craving in Response to the Alcohol Cue Script
Description: as for outcome 1
Time Frame: 15 minutes after the beginning of script presentation, which occurred on Day 21, 22, or 23 of the treatment period
Population: The analyses included only those subjects who completed all three script types (neutral, alcohol, stress)
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 6 | 8
Units on a scale | 17.4172 (2.3136) | 9.8121 (1.9853)

4. Primary Outcome: Alcohol Craving in Response to the Alcohol Cue Script
Description: as for outcome 1
Time Frame: 30 minutes after the beginning of script presentation, which occurred on Day 21, 22, or 23 of the treatment period
Population: The analyses included only those subjects who completed all three script types (neutral, alcohol, stress)
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 6 | 8
Units on a scale | 19.0838 (2.3136) | 10.5621 (1.9853)

5. Primary Outcome: Alcohol Craving in Response to the Alcohol Cue Script
Description: as for outcome 1
Time Frame: 45 minutes after the beginning of script presentation, which occurred on Day 21, 22, or 23 of the treatment period
Population: The analyses included only those subjects who completed all three script types (neutral, alcohol, stress)
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 6 | 8
Units on a scale | 18.0838 (2.3136) | 8.4371 (1.9853)

6. Primary Outcome: Alcohol Craving in Response to the Alcohol Cue Script
Description: as for outcome 1
Time Frame: 60 minutes after the beginning of script presentation, which occurred on Day 21, 22, or 23 of the treatment period
Population: The analyses included only those subjects who completed all three script types (neutral, alcohol, stress)
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 6 | 8
Units on a scale | 16.4172 (2.3136) | 8.9371 (1.9853)

7. Primary Outcome: Alcohol Craving in Response to the Alcohol Cue Script
Description: as for outcome 1
Time Frame: 75 minutes after the beginning of script presentation, which occurred on Day 21, 22, or 23 of the treatment period
Population: The analyses included only those subjects who completed all three script types (neutral, alcohol, stress)
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 6 | 8
Units on a scale | 15.2505 (2.3136) | 9.6871 (1.9853)

8. Primary Outcome: Alcohol Craving in Response to the Alcohol Cue Script
Description: as for outcome 1
Time Frame: 90 minutes after the beginning of script presentation, which occurred on Day 21, 22, or 23 of the treatment period
Population: The analyses included only those subjects who completed all three script types (neutral, alcohol, stress)
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 6 | 8
Units on a scale | 19.2505 (2.3136) | 8.9371 (1.9853)

9. Primary Outcome: Alcohol Craving in Response to the Lipopolysaccharide Challenge
Description: as for outcome 1
Time Frame: 15 minutes prior to the subject receiving an intravenous bolus of lipopolysaccharide, which occurred on Day 25 or Day 32 of the treatment period
Population: The analyses included only those subjects who completed both the lipopolysaccharide and placebo challenge sessions
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 5 | 8
Units on a scale | 11.1285 (1.5864) | 10.7947 (1.2432)

10. Primary Outcome: Alcohol Craving in Response to the Lipopolysaccharide Challenge
Description: as for outcome 1
Time Frame: 1 hour after the subject received an intravenous bolus of lipopolysaccharide, which occurred on Day 25 or Day 32 of the treatment period
Population: The analyses included only those subjects who completed both the lipopolysaccharide and placebo challenge sessions
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 5 | 8
Units on a scale | 9.5285 (1.5864) | 9.1697 (1.2432)

11. Primary Outcome: Alcohol Craving in Response to the Lipopolysaccharide Challenge
Description: as for outcome 1
Time Frame: 2 hours after the subject received an intravenous bolus of lipopolysaccharide, which occurred on Day 25 or Day 32 of the treatment period
Population: The analyses included only those subjects who completed both the lipopolysaccharide and placebo challenge sessions
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 5 | 8
Units on a scale | 11.9285 (1.5864) | 9.0447 (1.2432)

12. Primary Outcome: Alcohol Craving in Response to the Lipopolysaccharide Challenge
Description: as for outcome 1
Time Frame: 3 hours after the subject received an intravenous bolus of lipopolysaccharide, which occurred on Day 25 or Day 32 of the treatment period
Population: The analyses included only those subjects who completed both the lipopolysaccharide and placebo challenge sessions
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 5 | 8
Units on a scale | 9.5285 (1.5864) | 10.5447 (1.2432)

13. Primary Outcome: Alcohol Craving in Response to the Lipopolysaccharide Challenge
Description: as for outcome 1
Time Frame: 4 hours after the subject received an intravenous bolus of lipopolysaccharide, which occurred on Day 25 or Day 32 of the treatment period
Population: The analyses included only those subjects who completed both the lipopolysaccharide and placebo challenge sessions
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 5 | 8
Units on a scale | 12.1285 (1.5864) | 10.5447 (1.2432)

14. Primary Outcome: Alcohol Craving in Response to the Lipopolysaccharide Challenge
Description: as for outcome 1
Time Frame: 5 hours after the subject received an intravenous bolus of lipopolysaccharide, which occurred on Day 25 or Day 32 of the treatment period
Population: The analyses included only those subjects who completed both the lipopolysaccharide and placebo challenge sessions
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 5 | 8
Units on a scale | 12.1285 (1.5864) | 10.9197 (1.2432)

15. Primary Outcome: Alcohol Craving in Response to the Lipopolysaccharide Challenge
Description: as for outcome 1
Time Frame: 6 hours after the subject received an intravenous bolus of lipopolysaccharide, which occurred on Day 25 or Day 32 of the treatment period
Population: The analyses included only those subjects who completed both the lipopolysaccharide and placebo challenge sessions
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 5 | 8
Units on a scale | 9.9285 (1.5864) | 9.6697 (1.2432)

16. Primary Outcome: Alcohol Craving in Response to the Stress Script
Description: as for outcome 1
Time Frame: 15 minutes prior to the beginning of script presentation, which occurred on Day 21, 22, or 23 of the treatment period
Population: The analyses included only those subjects who completed all three script types (neutral, alcohol, stress)
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 6 | 8
Units on a scale | 10 (1.779) | 11.25 (1.5406)

17. Primary Outcome: Alcohol Craving in Response to the Stress Script
Description: as for outcome 1
Time Frame: 15 minutes after the beginning of script presentation, which occurred on Day 21, 22, or 23 of the treatment period
Population: The analyses included only those subjects who completed all three script types (neutral, alcohol, stress)
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 6 | 8
Units on a scale | 10 (1.779) | 12.125 (1.5406)

18. Primary Outcome: Alcohol Craving in Response to the Stress Script
Description: as for outcome 1
Time Frame: 5 minutes after the beginning of script presentation, which occurred on Day 21, 22, or 23 of the treatment period
Population: The analyses included only those subjects who completed all three script types (neutral, alcohol, stress)
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 6 | 8
Units on a scale | 10.3333 (1.779) | 11.875 (1.5406)

19. Primary Outcome: Alcohol Craving in Response to the Stress Script
Description: as for outcome 1
Time Frame: 30 minutes after the beginning of script presentation, which occurred on Day 21, 22, or 23 of the treatment period
Population: The analyses included only those subjects who completed all three script types (neutral, alcohol, stress)
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 6 | 8
Units on a scale | 10 (1.779) | 11.375 (1.5406)

20. Primary Outcome: Alcohol Craving in Response to the Stress Script
Description: as for outcome 1
Time Frame: 45 minutes after the beginning of script presentation, which occurred on Day 21, 22, or 23 of the treatment period
Population: The analyses included only those subjects who completed all three script types (neutral, alcohol, stress)
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 6 | 8
Units on a scale | 10.1667 (1.779) | 9.125 (1.5406)

21. Primary Outcome: Alcohol Craving in Response to the Stress Script
Description: as for outcome 1
Time Frame: 60 minutes after the beginning of script presentation, which occurred on Day 21, 22, or 23 of the treatment period
Population: The analyses included only those subjects who completed all three script types (neutral, alcohol, stress)
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 6 | 8
Units on a scale | 10.1667 (1.779) | 9.25 (1.5406)

22. Primary Outcome: Alcohol Craving in Response to the Stress Script
Description: as for outcome 1
Time Frame: 75 minutes after the beginning of script presentation, which occurred on Day 21, 22, or 23 of the treatment period
Population: The analyses included only those subjects who completed all three script types (neutral, alcohol, stress)
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 6 | 8
Units on a scale | 10.1667 (1.779) | 9.5 (1.5406)

23. Primary Outcome: Alcohol Craving in Response to the Stress Script
Description: as for outcome 1
Time Frame: 90 minutes after the beginning of script presentation, which occurred on Day 21, 22, or 23 of the treatment period
Population: The analyses included only those subjects who completed all three script types (neutral, alcohol, stress)
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 6 | 8
Units on a scale | 10.6667 (1.779) | 9.625 (1.5406)

24. Secondary Outcome: Anxiety Symptom Ratings Measured Bi-weekly During the Treatment Period
Description: Anxiety symptoms were measured using the Comprehensive Psychopathological Rating Scale (CPRS). The CPRS is an 18-item interview-based instrument for assessing depression and anxiety. There are two 10-item subscales, the Montgomery-Asberg Depression Rating Scale (MADRS) and the Brief Scale for Anxiety (BSA). Each subscale ranges from 0 (lowest symptom severity) to 60 (highest symptom severity).
Time Frame: Day 1 of the treatment period
Population: The analyses included only those subjects who had a baseline anxiety symptom rating taken 1 day after inpatient admission (but prior to enrollment in this protocol), and who completed all 33 days of the treatment period
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 6 | 8
Units on a scale | 2.8502 (1.4379) | 4.5791 (1.235)

25. Secondary Outcome: Anxiety Symptom Ratings Measured Bi-weekly During the Treatment Period
Description: as for outcome 24
Time Frame: Day 3 of the treatment period
Population: as for outcome 24
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 6 | 8
Units on a scale | 5.884 (1.3775) | 0.5706 (1.1885)

26. Secondary Outcome: Anxiety Symptom Ratings Measured Bi-weekly During the Treatment Period
Description: as for outcome 24
Time Frame: Day 7 of the treatment period
Population: as for outcome 24
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 6 | 8
Units on a scale | 3.2897 (1.4413) | 2.0706 (1.1885)

27. Secondary Outcome: Anxiety Symptom Ratings Measured Bi-weekly During the Treatment Period
Description: as for outcome 24
Time Frame: Day 10 of the treatment period
Population: as for outcome 24
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 6 | 8
Units on a scale | 3.3403 (1.4413) | 1.1956 (1.1885)

28. Secondary Outcome: Anxiety Symptom Ratings Measured Bi-weekly During the Treatment Period
Description: as for outcome 24
Time Frame: Day 14 of the treatment period
Population: as for outcome 24
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 6 | 8
Units on a scale | 4.2173 (1.3775) | 1.2136 (1.2176)

29. Secondary Outcome: Anxiety Symptom Ratings Measured Bi-weekly During the Treatment Period
Description: as for outcome 24
Time Frame: Day 17 of the treatment period
Population: as for outcome 24
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 6 | 8
Units on a scale | 5.0507 (1.3775) | 1.0706 (1.1885)

30. Secondary Outcome: Anxiety Symptom Ratings Measured Bi-weekly During the Treatment Period
Description: as for outcome 24
Time Frame: Day 21 of the treatment period
Population: as for outcome 24
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 6 | 8
Units on a scale | 5.0507 (1.3775) | 1.6956 (1.1885)

31. Secondary Outcome: Anxiety Symptom Ratings Measured Bi-weekly During the Treatment Period
Description: as for outcome 24
Time Frame: Day 24 of the treatment period
Population: as for outcome 24
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 6 | 8
Units on a scale | 3.884 (1.3775) | 0.6956 (1.1885)

32. Secondary Outcome: Anxiety Symptom Ratings Measured Bi-weekly During the Treatment Period
Description: as for outcome 24
Time Frame: Day 28 of the treatment period
Population: as for outcome 24
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 6 | 8
Units on a scale | 4.884 (1.3775) | 1.1125 (1.2543)

33. Secondary Outcome: Anxiety Symptom Ratings Measured Bi-weekly During the Treatment Period
Description: as for outcome 24
Time Frame: Day 31 of the treatment period
Population: as for outcome 24
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 6 | 8
Units on a scale | 7.2173 (1.3775) | 1.8206 (1.1885)

34. Secondary Outcome: Depression Symptom Ratings Measured Bi-weekly During the Treatment Period
Description: Depression symptoms were measured using the Comprehensive Psychopathological Rating Scale (CPRS). The CPRS is an 18-item interview-based instrument for assessing depression and anxiety. There are two 10-item subscales, the Montgomery-Asberg Depression Rating Scale (MADRS) and the Brief Scale for Anxiety (BSA). Each subscale ranges from 0 (lowest symptom severity) to 60 (highest symptom severity).
Time Frame: Day 1 of the treatment period
Population: The analyses included only those subjects who had a baseline depression symptom rating taken 1 day after inpatient admission (but prior to enrollment in this protocol), and who completed all 33 days of the treatment period
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 6 | 8
Units on a scale | 6.3661 (1.4855) | 3.2956 (1.275)

35. Secondary Outcome: Depression Symptom Ratings Measured Bi-weekly During the Treatment Period
Description: as for outcome 34
Time Frame: Day 3 of the treatment period
Population: as for outcome 34
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 6 | 8
Units on a scale | 5.6366 (1.4174) | 0.9937 (1.2232)

36. Secondary Outcome: Depression Symptom Ratings Measured Bi-weekly During the Treatment Period
Description: as for outcome 34
Time Frame: Day 7 of the treatment period
Population: as for outcome 34
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 6 | 8
Units on a scale | 4.9065 (1.4906) | 0.9937 (1.2232)

37. Secondary Outcome: Depression Symptom Ratings Measured Bi-weekly During the Treatment Period
Description: as for outcome 34
Time Frame: Day 10 of the treatment period
Population: as for outcome 34
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 6 | 8
Units on a scale | 4.7167 (1.4906) | 0.8687 (1.2232)

38. Secondary Outcome: Depression Symptom Ratings Measured Bi-weekly During the Treatment Period
Description: as for outcome 34
Time Frame: Day 14 of the treatment period
Population: as for outcome 34
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 6 | 8
Units on a scale | 4.6366 (1.4174) | 0.5912 (1.2569)

39. Secondary Outcome: Depression Symptom Ratings Measured Bi-weekly During the Treatment Period
Description: as for outcome 34
Time Frame: Day 17 of the treatment period
Population: as for outcome 34
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 6 | 8
Units on a scale | 6.3032 (1.4174) | 0.8687 (1.2232)

40. Secondary Outcome: Depression Symptom Ratings Measured Bi-weekly During the Treatment Period
Description: as for outcome 34
Time Frame: Day 21 of the treatment period
Population: as for outcome 34
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 6 | 8
Units on a scale | 5.1366 (1.4174) | 1.4937 (1.2232)

41. Secondary Outcome: Depression Symptom Ratings Measured Bi-weekly During the Treatment Period
Description: as for outcome 34
Time Frame: Day 24 of the treatment period
Population: as for outcome 34
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 6 | 8
Units on a scale | 7.1366 (1.4174) | 1.1187 (1.2232)

42. Secondary Outcome: Depression Symptom Ratings Measured Bi-weekly During the Treatment Period
Description: as for outcome 34
Time Frame: Day 28 of the treatment period
Population: as for outcome 34
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 6 | 8
Units on a scale | 6.4699 (1.4174) | 1.1228 (1.299)

43. Secondary Outcome: Depression Symptom Ratings Measured Bi-weekly During the Treatment Period
Description: as for outcome 34
Time Frame: Day 31 of the treatment period
Population: as for outcome 34
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 6 | 8
Units on a scale | 8.6366 (1.4174) | 0.8687 (1.2232)

44. Secondary Outcome: Spontaneous Alcohol Craving Measured Bi-weekly During the Treatment Period
Description: Alcohol craving was measured using the Penn Alcohol Craving Scale (PACS). The PACS is a five-item self-administered instrument for assessing alcohol craving over the course of the past week. The score ranges from 0 (lowest craving value) to 30 (highest craving value).
Time Frame: Day 1 of the treatment period
Population: The analyses included only those subjects who had a baseline craving measure taken 4 days after inpatient admission (but prior to enrollment in this protocol), and who completed all 33 days of the treatment period
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 6 | 8
Units on a scale | 7.7503 (1.7317) | 7.8122 (1.4976)

45. Secondary Outcome: Spontaneous Alcohol Craving Measured Bi-weekly During the Treatment Period
Description: as for outcome 44
Time Frame: Day 3 of the treatment period
Population: as for outcome 44
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 6 | 8
Units on a scale | 8.417 (1.7317) | 5.9372 (1.4976)

46. Secondary Outcome: Spontaneous Alcohol Craving Measured Bi-weekly During the Treatment Period
Description: as for outcome 44
Time Frame: Day 7 of the treatment period
Population: as for outcome 44
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 6 | 8
Units on a scale | 7.0837 (1.7317) | 4.1872 (1.4976)

47. Secondary Outcome: Spontaneous Alcohol Craving Measured Bi-weekly During the Treatment Period
Description: as for outcome 44
Time Frame: Day 10 of the treatment period
Population: as for outcome 44
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 6 | 8
Units on a scale | 6.0837 (1.7317) | 3.9372 (1.4976)

48. Secondary Outcome: Spontaneous Alcohol Craving Measured Bi-weekly During the Treatment Period
Description: as for outcome 44
Time Frame: Day 14 of the treatment period
Population: as for outcome 44
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 6 | 8
Units on a scale | 4.7503 (1.7317) | 4.1872 (1.4976)

49. Secondary Outcome: Spontaneous Alcohol Craving Measured Bi-weekly During the Treatment Period
Description: as for outcome 44
Time Frame: Day 17 of the treatment period
Population: as for outcome 44
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 6 | 8
Units on a scale | 4.7503 (1.7317) | 4.0622 (1.4976)

50. Secondary Outcome: Spontaneous Alcohol Craving Measured Bi-weekly During the Treatment Period
Description: as for outcome 44
Time Frame: Day 21 of the treatment period
Population: as for outcome 44
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 6 | 8
Units on a scale | 4.417 (1.7317) | 3.8122 (1.4976)

51. Secondary Outcome: Spontaneous Alcohol Craving Measured Bi-weekly During the Treatment Period
Description: as for outcome 44
Time Frame: Day 24 of the treatment period
Population: as for outcome 44
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 6 | 8
Units on a scale | 5.917 (1.7317) | 2.3122 (1.4976)

52. Secondary Outcome: Spontaneous Alcohol Craving Measured Bi-weekly During the Treatment Period
Description: as for outcome 44
Time Frame: Day 28 of the treatment period
Population: as for outcome 44
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 6 | 8
Units on a scale | 6.417 (1.7317) | 2.6872 (1.4976)

53. Secondary Outcome: Spontaneous Alcohol Craving Measured Bi-weekly During the Treatment Period
Description: as for outcome 44
Time Frame: Day 31 of the treatment period
Population: as for outcome 44
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 6 | 8
Units on a scale | 4.5837 (1.7317) | 2.8122 (1.4976)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected throughout the 31 days of the inpatient stay for each subject
Arm/Group | Pioglitazone | Placebo
Serious Adverse Events (participants affected / at risk) | 2/8 | 0/8
Other Adverse Events (participants affected / at risk) | 8/8 | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pioglitazone (N=8) | Placebo (N=8)
Abnormal glucose (Investigations) | 1 | 0
Elevated Creatine Kinase (Investigations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pioglitazone (N=8) | Placebo (N=8)
Blurred vision (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Bloating (Gastrointestinal disorders) | 1 | 0
Blood in stool (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 2
Stomach pain (Gastrointestinal disorders) | 1 | 1
Toothache (Gastrointestinal disorders) | 1 | 3
Buzzed (General disorders) | 1 | 0
Chills (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Fever (General disorders) | 1 | 0
Irritability (General disorders) | 0 | 1
Loss of Appetite (General disorders) | 2 | 0
Low RBC/HGB A1C (General disorders) | 1 | 0
Pain (General disorders) | 2 | 0
Sleepiness (General disorders) | 1 | 1
Tiredness (General disorders) | 5 | 5
Trouble Sleeping (General disorders) | 1 | 0
Abnormal platelet count (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Elevated Creatine Kinase (Investigations) | 4 | 1
Muscle aches (Musculoskeletal and connective tissue disorders) | 1 | 3
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 4
Light headed (Nervous system disorders) | 1 | 1
Sinus pain (Nervous system disorders) | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 1
Dark Urine (Renal and urinary disorders) | 0 | 1
Urinary frequency (Renal and urinary disorders) | 0 | 1
Cold-like symptoms (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Acne (Skin and subcutaneous tissue disorders) | 0 | 1
Itching (Skin and subcutaneous tissue disorders) | 1 | 1
Phlebitis (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
This study was terminated early, so the number of subjects analyzed is small.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes